CLINICAL TRIAL: NCT05903781
Title: Value of Ultra-fast Biparametric MRI in the Assessment of Prostate Cancer
Brief Title: Value of Ultra-fast Prostate MRI in Prostate Cancer
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: Ultra- Fast Prostate MRI
Record Dates: First submitted 2023-05-31; First posted 2023-06-15 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Prostate MRI — MRI of the prostate

SUMMARY:
This study aims to assess the value of ultra-fast MRI sequences in the assessment of prostate cancer, compared to the full multiparametric/biparametric protocol as the clinical standard.

DETAILED DESCRIPTION:
Prostate cancer is the second most common type of cancer among men and the fifth leading cause of cancer-related deaths globally. Magnetic resonance imaging (MRI) has become an integral part of the clinical assessment of prostate cancer and is a valuable tool to identify target lesions for subsequent biopsy, perform local tumor staging, provide information on active surveillance approaches, and might also be eligible for prostate cancer screening.

To standardize the interpretation and reporting in prostate MRI, the PI-RADS (Prostate Imaging-Reporting and Data System) scoring system has been developed. PI-RADS has played a crucial role in the widespread adoption of prostate MRI among radiologists and urologists worldwide and has also become an essential part of national and international clinical guidelines. This has resulted in a notable surge in the number of prostate MRI examinations conducted in recent years, and is expected to further increase over the next years. The present PI-RADS guideline provides comprehensive technical instructions on the acquisition of prostate MRI leading to the acquisition of a multiparametric MRI (mpMRI) that typically requires around 30 minutes of scan time.

As healthcare systems around the world face increasing demand and limited resources, there is a need to identify efficient and cost-effective ways to diagnose and treat prostate cancer. Efforts have been made to reduce the duration and expenses associated with prostate MRI acquisition and interpretation, leading to a biparametric MRI (bpMRI, exclusion of contrast-enhanced sequences) with a shortened protocol compared to the conventional mpMRI. Several studies have demonstrated the high diagnostic accuracy of abbreviated prostate MRI for detecting and even staging prostate cancer in comparison to traditional full mpMRI. The accelerated protocols have therefore the potential to improve efficiency and patient comfort, to reduce healthcare costs and make this technique accessible to more men. Nevertheless, even these shortened protocols accrue a scan time of about 15-20 minutes. Recent developments in MRI technique now allow for even faster image acquisitions, but more research is necessary to fully elicit the advantages and limitations of accelerated or even ultra-fast prostate MRI protocols (scan time of < 5 min) before incorporating them into routine clinical practice.

The purpose of this study is therefore to further explore ultra-fast bpMRI compared to conventional full mpMRI of the prostate to gain valuable insights into the diagnostic performance, feasibility and clinical utility of this emerging imaging technique and consequently optimize prostate cancer management.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo clinically indicated MR imaging of the prostate
* Informed consent as documented by signature (Informed Consent Form)
* Patients ≥18 years of age

Exclusion Criteria:

* Inability to follow the procedures of the study, e.g., due to language problems, psychological disorders, dementia, etc. of the participant
* Previous enrolment into the current study
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* Patients with non-MRI compatible metallic or electronic implants, devices or metallic foreign bodies (cardiac pacemaker, shrapnel, cochlea implants, neurostimulator, or other non-MRI compatible implants).
* Patients with known hypersensitivity reactions to MRI contrast agents will undergo the examination without application of a contrast agent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ca. 300 men with suspected prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 536 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2025-02-18 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of ultrafast bpMRI of the prostate | 1.5 years
  Diagnostic accuracy of ultrafast bpMRI of the prostate

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No